CLINICAL TRIAL: NCT03224832
Title: Pancreatoduodenectomy With Mesopancreas Dissection.A Prospective Study Comparing Artery-first Approach Versus Standard Approach
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Moustafa Ali Sayed Mahmoud, Assistant lecturer at General surgery department, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: mas2017
Record Dates: First submitted 2017-07-13; First posted 2017-07-21 (Actual); Last update posted 2017-08-10 (Actual); Status verified 2017-05

CONDITIONS: Periampullary Carcinoma Resectable

STUDY DESIGN:
Intervention Model Description: one group will be subjected to artery fgirst approach at EL Rajhi hospital and the other group will be subjected to standard approach at the main general surgery department at Assiut university hospital
Who Masked: Participant
Masking Description: the cases which will come to general surgery outpatient clinic will be subjected to standard approach while the cases which will come to our EL Rajhi outpatient clinic will be subjected to artery-first approach
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group 1 (Experimental): group 1 will be Pancreatoduodenectomy With Mesopancreas. Artery-first Approach
  Interventions: Procedure: Artery-first Approach
- group2 (Experimental): group2 will be Pancreatoduodenectomy With Mesopancreas Dissection. Standard Approach
  Interventions: Procedure: Standard Approach

INTERVENTIONS:
Procedure: Artery-first Approach — Dissection at the origin of the superior mesenteric artery and the celiac trunk all along their right side of the vessels. -En bloc resection of the primary tumor and regional lymph nodes through complete excision of the mesopancreatic plane, utilizing the artery-first approach.
  * The mesopancreatic plane consists of the pancreas head, the uncinate process of the pancreas, and the meso-pancreatoduodenum.
  All the tissues that lay in this triangular space (SMA down, CT up, and SMV-PV anterior) is cleared.
  Then the investigators continue the dissection along the right then anterior surface of the SMV and PV until reaching the dissected posterior surface the neck of the pancreas .
  Last step is the division of the neck of the pancreas. After the specimen is removed and before it is sent to the pathology we put mark on each boundary of the specimen one towards SMA, another towards PV/SMV area and the last towards the posterior surface of the mesopancreas.
  Other Names: group 1
  Arms: group 1
Procedure: Standard Approach — In standard approach after kocharization of the duodenum the investigators start to asses the tunnel under the neck of the pancreas whether tumor infilterating PV/SMV axis and if not we cut the neck of pancreas early in the procedure then we continue to dissect the uncinate process and control pancreatoduodenal vessels and draining lymph nodes and LNS around portal vein and up to hepatic artery and we will add to the standard procedure the previously defined mesopancreatic triangle dissection which lies between SMA caudal, Coeliac artery cranial and PV/SMV axis anterior and the specimen will be marked and sent as previous to pathology.
  Other Names: group2
  Arms: group2

SUMMARY:
The definitions for R0 and R1 margin status after resection for pancreatic cancer are controversial.Various studies showed the rate of noncurative resections of 15- 35 % but with modified pathological examination (R1/R2) revealed the rate of R1 resection was higher ranging from 76-85 % .

Verbeke CS etal.

* Whether this discrepancy was caused by incomplete lymphnode dissection, perineural dissection and improper pathological examination was not yet known.
* Perineural invasion was detected in 77 % of specimens of resected pancreatic cancers.

So the researchers emphasized the need of new surgical classification involving mesopancreas. It can be considered as an anatomical space bounded anteriorly by the the posterior surface of the pancreatic neck, posteriorly by the pancreaticoduodenal coalescence fascia, medially by the mesenteric vessels with -nerves, lymphatics and vessels as its contents.

DETAILED DESCRIPTION:
A Controlled clinical trial of pancreatoduodenectomy with mesopancreas dissection.A Prospective study comparing artery-first versus standard approach.

* Target population:

  -All cases of malignant obstructive jaundice within the above criteria.
* Sample size:

  * It will be conventional sample size of about 40 cases minimum about 20 case for each group of the both procedures
  * Techniques:
  * The procedure at Assiut university hospital consists of artery-first with l dissection at the origin of the superior mesenteric artery and the celiac trunk all along their right side of the vessels versus standard approach.
  * This allows a complete clearance of retro- pancreatic tissues.
  * -En bloc resection of the primary tumor and regional lymph nodes through complete excision of the mesopancreatic plane, utilizing the artery-first approach.
  * -The mesopancreatic plane consists of the pancreas head, the uncinate process of the pancreas, and the meso-pancreatoduodenum.
  * All the tissues that lay in this triangular space (SMA down, CT up, and SMV-PV anterior) is cleared.

Then the investigators continue the dissection along the right then anterior surface of the SMV and PV until reaching the dissected posterior surface the neck of the pancreas .

* Last step is the division of the neck of the pancreas.
* After the specimen is removed and before it is sent to the pathology the investigators put mark on each boundary of the specimen one towards SMA, another towards PV/SMV area and the last towards the posterior surface of the mesopancreas.
* This can guide the pathologist to identify the retro pancreatic margins and define whenever there is an R1 resection the exact area of invasion. Microscopic margin involvement (R1) will be defined as tumor within 1 mm of resection margin.

While in standard approach at first kocharization of the duodenum ,then starting to asses the tunnel under the neck of the pancreas whether tumor infilterating PV/SMV axis and if not the investigators cut the neck of pancreas early in the procedure then continue to dissect the uncinate process and control pancreatoduodenal vessels and draining lymph nodes and LNS around portal vein and up to hepatic artery and we will add to the standard procedure the previously defined mesopancreatic triangle dissection which lies between SMA caudal, Coeliac artery cranial and PV/SMV axis anterior and the specimen will be marked and sent as previous to pathology.

ELIGIBILITY:
Inclusion Criteria:

* All cases of resectable periampullary carcinoma
* surgically fit accordying to ASA

Exclusion Criteria:

* Surgically unfit cases according to ASA.
* locally advanced irresectable cases

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-08 (Estimated); Primary Completion 2019-07-01 (Estimated); Study Completion 2020-01-01 (Estimated)

PRIMARY OUTCOMES:
Time to judge resectability intra operative and operative time for each procedure. | up to 2 weeks postoperative data will be available
  Time to judge resectability intra operative and operative time for each procedure usually lasts from 3 to 12 hours(operative time)
Blood loss in both procedures. | up to 2 weeks postoperative data will be available
  Blood loss in both procedures in cc usually lasts from 3 to 12 hours(operative time)
Pathological data | up to 2 weeks postoperative data will be available
  ( cancer type, grade,LNS number and focus on infiltration of mesopancreas(R0 free margin more than 1 mm R1 +margin or infiltration less than 1mm.
Mortality rate. | up to 15 months after each case
  number of deaths intraoperative and immediate postoperative

SECONDARY OUTCOMES:
- Short term postoperative survival 15 month after the last case of the study | 15 month after the last case of the study
  - Short term postoperative survival 15 month after the last case of the study
locoregional recurrence | 15 month after the last case of the study
  locoregional recurrence follow up ct abdomen every 4 months postoperative till 15 months postoperative
Postoperative complications | 15 month after the last case of the study
  Postoperative complications especially diarrhea

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
Prospective comparative study between Artery-first versus standard pancreatoduodenectomy with mesopancreas dissection.
  Evaluating perioperative outcomes:Blood loss,Operative time(+/-time to judge resectability),Pathological data(specially those related to mesopancreas) morbidity and mortality

REFERENCES:
- [Result] Adham M, Singhirunnusorn J. Surgical technique and results of total mesopancreas excision (TMpE) in pancreatic tumors. Eur J Surg Oncol. 2012 Apr;38(4):340-5. doi: 10.1016/j.ejso.2011.12.015. Epub 2012 Jan 20. PMID 22264964
- [Result] Kayahara M, Nagakawa T, Ueno K, Ohta T, Takeda T, Miyazaki I. An evaluation of radical resection for pancreatic cancer based on the mode of recurrence as determined by autopsy and diagnostic imaging. Cancer. 1993 Oct 1;72(7):2118-23. doi: 10.1002/1097-0142(19931001)72:73.0.co;2-4. PMID 8104092
- [Result] Gockel I, Domeyer M, Wolloscheck T, Konerding MA, Junginger T. Resection of the mesopancreas (RMP): a new surgical classification of a known anatomical space. World J Surg Oncol. 2007 Apr 25;5:44. doi: 10.1186/1477-7819-5-44. PMID 17459163
- See also: Clearance of the retropancreatic margin in pancreatic carcinomas: total mesopancreas excision or extended lymphadenectomy? [Eur J Surg Oncol. 2012] — https://www.ncbi.nlm.nih.gov/pubmed/?term=Surgical+technique+and+results+of+total+mesopancreas+excision+(TMpE)+in+pancreatic+tumors
- See also: The frequency of retroperitoneal recurrence of carcinoma of the head of the pancreas suggests that retroperitoneal resection, — https://www.ncbi.nlm.nih.gov/pubmed/?term=)+An+evaluation+of+radical+resection+for+pancreatic+cancer+based+on+the+mode+of+recurrence+as+determined+by+autopsy+and+diagnostic+imaging
- See also: The aim to ensure the greatest possible distance from the retropancreatic lymphatic tissue which drains the carcinomatous focus can be achieved in patients with pancreatic cancer only by complete resection of the mesopancreas (RMP). — http://www.ncbi.nlm.nih.gov/pubmed/?term=Resection+of+the+mesopancreas+(RMP)%3A+a+new+surgical+classification+of+a+known+anatomical+space